CLINICAL TRIAL: NCT03165513
Title: Dialogue to Empower, Supervise, Support and Include the Traditional and Faith Healers to Deliver Evidence-based mhGAP-IG Adapted Psychosocial Interventions to Reduce Treatment Gap in Kenya
Brief Title: Dialogue to Empower Traditional and Faith Healers to Deliver mhGAP-IG Adapted Psychosocial Interventions in Kenya
Acronym: Dialogue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P602/12/2013
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Depressive Disorder, Major
Keywords: Traditional healer; faith healer; depression; mhGAP; Kenya
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): mhGAP-IG psychosocial intervention
  Interventions: Behavioral: mhGAP-IG

INTERVENTIONS:
Behavioral: mhGAP-IG — psychosocial interventions

SUMMARY:
The project aimed to create a dialogue between the informal sector (traditional and faith healers) and the formal sector (trained health care workers) in order to increase synergy and communication between the two systems, by minimizing any harmful practices and enhancing complementary practices. The informal sector will also be trained on how to use WHO mhGAP-IG component on depression for routine screening in order to ameliorate functional and social outcomes and refer complicated cases to the formal sector for biological interventions

DETAILED DESCRIPTION:
This study seeks to empower, supervise, support and include the informal traditional and faith healers to deliver evidence-based mhGAP-IG adapted psychosocial interventions to reduce mental health treatment gap in Kenya. This will be achieved through establishing a dialogue and collaboration between the formal and the informal sector and training the informal sector on the use of mental health Gap Action Programme Intervention Guideline (mhGAP-IG) to identify and manage depression. It will take place in Makueni County among 100 randomly selected TH/FH. A descriptive (prospective cohort) study will be used to determine the impact of training TH/FH on the use of mhGAP-IG in the identification and management of depression. A mental health specialist will also determine the accuracy of diagnosis made by the informal sector using randomly selected patients (true positives and true negatives for depression) by an independent person. Moreover, patients identified to have depression will be followed up at 6 and 12 weeks to assess their health outcomes using BECKs Depression Inventory Scale, Suicidality Scale and WHO quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Traditional and faith healers residing in Kibwezi West constituency
2. Traditional and faith healers who are willing to participate in the study.
3. Traditional and faith healers' patients' above 18 years who agree to participate in the study

Exclusion Criteria:

1. Traditional and faith healers not residing in Kibwezi West constituency
2. Traditional and faith healers who are not willing to participate in the study.
3. Traditional and faith healers' patients' above 18 years who do not agree to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4081 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Depression symptoms on the Becks Depression Inventory Scale | Baseline, 6 weeks and 12 weeks
  Changes in depression scores (over time) on the Becks Depression Inventory Scale

SECONDARY OUTCOMES:
Quality of life outcomes on the WHO Quality of Life-BREF (WHOQOL-BREF) | baseline, 6 weeks and 12 weeks
  Changes in quality of life domains using WHO Quality of Life-BREF (WHOQOL-BREF)

CONTACTS AND LOCATIONS:
Overall Officials: Christine W Musyimi, MSc, Principal Investigator — Africa Institute of Mental and Brain Health (AFRIMEB)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available to the researchers on request through the principal investigator. A data request form available at AMHF will be used to make the request

REFERENCES:
- See also: Forming a joint dialogue article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4705751/
- See also: Mental Health Outcomes of Psychosocial Intervention Among Traditional Health Practitioner Depressed Patients in Kenya. — https://www.ncbi.nlm.nih.gov/pubmed/28251478
- See also: Quality of life of depressed and suicidal patients seeking services from traditional and faith healers in rural Kenya — https://www.ncbi.nlm.nih.gov/pubmed/28482849